CLINICAL TRIAL: NCT04787978
Title: Creating Healthier Communities Through Meaningful Partnerships: A Model From the National African American Male Wellness Initiative - OSU Partnership
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Joshua Joseph, MD, Assistant Professor of Medicine, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019H0302
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Hypertension; Diabetes; Sedentary Behavior; High Cholesterol; Diet, Healthy; Smoking Reduction; Weight Loss
MeSH Terms: conditions — Hypertension; Diabetes Mellitus; Sedentary Behavior; Hypercholesterolemia; Smoking Reduction; Weight Loss | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: single-arm pilot program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AAMWI-OSU Intervention (Experimental): In this single-arm pilot program, 100 African American male participants will be enrolled who have poor or average cardiovascular health (< 4 life's simple 7 metrics in the ideal range) to a physical activity, education and patient activation intervention.
  Interventions: Other: Physical Activity and Education Intervention

INTERVENTIONS:
Other: Physical Activity and Education Intervention — The intervention involves peer teams, health coaches and community health workers [CHW]. Each participant will be assigned to a CHW and grouped into a team of 10-20 participants based on participant proximity to a Columbus Recreation and Parks Center. Each team will be assigned 4 health coaches, 2 medical students, 1 undergraduate student and 1 nursing student from OSU Health Sciences Colleges.
  The lifestyle intervention is 24 weeks consisting of 1 hour and 15 minutes of in person training time per week. The training time consists of 45 minutes of physical activity and 30 minutes of educational content was informed by evidence-based strategies and stakeholder feedback.
  Health coaches will implement the curriculum based on the Diabetes Prevention Program and the American Heart Association Check, Change, Control Program and develop team-based SMART (specific, measurable, achievable, relevant, and time-bound) wellness goals.

SUMMARY:
Primary Objective: Test feasibility and acceptability of a 24-week community-based lifestyle intervention to improve cardiovascular health among African American males.

Secondary Objectives: 1) Navigate participants to establish primary care and address social and patient activation needs that present barriers to wellness; 2) Examine changes in cardiovascular health as per American Heart Association Life's Simple 7 Metrics including blood pressure, cholesterol, glucose, smoking, body mass index, physical activity and dietary intake (1); and 3) Increase African American male participation in clinical trials.

DETAILED DESCRIPTION:
Chronic diseases, particularly diabetes (DM), cardiovascular disease (CVD), and cancer, pose a tremendous burden for Ohio residents, health systems, and employers. This burden is not equally distributed and mortality from these diseases is greatest among African American (AA) men. The National African American Male Wellness Initiative (AAMWI) was established in Columbus, Ohio in 2004. Through numerous events including an annual walk with health fair, the AAMWI aims to reduce premature mortality among AA males. It has become the largest health initiative in Central Ohio for AA's, spanning 5 cities in Ohio and total of 16 nationally. The Ohio State University (OSU) partners with the AAMWI to advance health equity in DM, CVD, and cancer. Through our partnership, community health workers (CHWs) and health coaches (HCs) aim to activate at-risk AA men to embrace wellness by: 1) facilitating engagement with a primary care provider and addressing social determinants of health that present barriers to wellness; 2) improving participants' "Life's Simple 7" (LS7) American Heart Association (AHA) metrics (blood pressure, cholesterol, glucose, smoking, body mass index, physical activity and dietary intake) through a community team-based intervention (Lloyd-Jones, 2010); and 3) increasing participation in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* African American men (self-report)
* Adult age 18 years or older
* Poor or average cardiovascular health (< 4 LS7 metrics in the ideal range) from the American Heart Association 2020 Guidelines
* Participant is appropriate for group setting.

Exclusion Criteria:

* Non-English speaking
* Living outside of the Metro Columbus Area
* Unable to perform physical activity

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2020-02-29 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-09-06 (Actual)

PRIMARY OUTCOMES:
Feasibility of a 24-week community-based lifestyle intervention to improve cardiovascular health among African American males | Week 1
  Feasibility, as assessed via enrollment, will be measured using the baseline study procedure logs.
Feasibility of a 24-week community-based lifestyle intervention to improve cardiovascular health among African American males | 24 weeks
  Feasibility, as assessed via retention, will be measured using attendance in the study procedure logs over the course of the study.
Acceptability of a 24-week community-based lifestyle intervention to change cardiovascular health among African American males | 24 weeks
  Protocol acceptability (satisfaction, usefulness, plans and change of behavior to apply health promotion strategies) will be assessed via structured questions in focus groups including satisfaction, usefulness and attainment of self-identified Specific, Measurable, Attainable, Relevant and Time-Based (SMART) goals.
Change in cardiovascular health (a composite measure of blood pressure, cholesterol, glucose, physical activity, smoking status, and body mass index). | 24 weeks
  Cardiovascular health will be assessed with seven metrics: smoking status, diet (Diet Health Questionnaire-III), physical activity (International Physical Activity Questionnaire), body mass index (kg/m2), serum cholesterol (mg/dl) and blood pressure (mmHg) and fasting glucose (mg/dl). Each baseline metric will be scored and categorized as poor, intermediate or ideal, as specified by AHA recommendations, with consideration of medication use (i.e. antihypertensive, lipid-lowering, glucose-lowering) where appropriate (Lloyd-Jones et al, 2010).
  Points will be allocated for each of the seven baseline metrics with scores of 0 poor, 1 intermediate or 2 ideal with a total score ranging from 0-14. Change in this score over 24 weeks will be examined (Joseph et al, 2016).

SECONDARY OUTCOMES:
Change in cardiovascular health (blood pressure, cholesterol, glucose, physical activity, smoking status, and body mass index as a composite measure (1,2)). | 12 weeks
  Cardiovascular health will be assessed with seven metrics: smoking status, diet (Diet Health Questionnaire-III), physical activity (International Physical Activity Questionnaire), body mass index (kg/m2), serum cholesterol (mg/dl) and blood pressure (mmHg) and fasting glucose (mg/dl). Each baseline metric will be scored and categorized as poor, intermediate or ideal, as specified by AHA recommendations, with consideration of medication use (i.e. antihypertensive, lipid-lowering, glucose-lowering) where appropriate (Lloyd-Jones et al, 2010).
  Points will be allocated for each of the seven baseline metrics with scores of 0 poor, 1 intermediate or 2 ideal with a total score ranging from 0-14. Change in this score over 12 weeks will be examined (Joseph et al, 2016).
Proportion of Participants with a Primary Care Provider | 24 weeks
  The change in proportion of participants with a primary care provider will be examined from 0 to 24 weeks.
Change in Patient Activation | 24 weeks
  Change in Insignia Health Patient Activation Measure will be examined from 0 to 24 weeks (Hibbard et al, 2004).

CONTACTS AND LOCATIONS:
Overall Officials: Darrell Gray, MD, Study Director — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lloyd-Jones DM, Hong Y, Labarthe D, Mozaffarian D, Appel LJ, Van Horn L, Greenlund K, Daniels S, Nichol G, Tomaselli GF, Arnett DK, Fonarow GC, Ho PM, Lauer MS, Masoudi FA, Robertson RM, Roger V, Schwamm LH, Sorlie P, Yancy CW, Rosamond WD; American Heart Association Strategic Planning Task Force and Statistics Committee. Defining and setting national goals for cardiovascular health promotion and disease reduction: the American Heart Association's strategic Impact Goal through 2020 and beyond. Circulation. 2010 Feb 2;121(4):586-613. doi: 10.1161/CIRCULATIONAHA.109.192703. Epub 2010 Jan 20. PMID 20089546
- [Background] Joseph JJ, Echouffo-Tcheugui JB, Carnethon MR, Bertoni AG, Shay CM, Ahmed HM, Blumenthal RS, Cushman M, Golden SH. The association of ideal cardiovascular health with incident type 2 diabetes mellitus: the Multi-Ethnic Study of Atherosclerosis. Diabetologia. 2016 Sep;59(9):1893-903. doi: 10.1007/s00125-016-4003-7. Epub 2016 Jun 8. PMID 27272340
- [Background] Hibbard JH, Stockard J, Mahoney ER, Tusler M. Development of the Patient Activation Measure (PAM): conceptualizing and measuring activation in patients and consumers. Health Serv Res. 2004 Aug;39(4 Pt 1):1005-26. doi: 10.1111/j.1475-6773.2004.00269.x. PMID 15230939
- [Derived] Joseph JJ, Nolan TS, Brock G, Williams A, Zhao S, McKoy A, Kluwe B, Metlock F, Campanelli K, Odei JB, Khumalo MT, Lavender D, Gregory J, Gray DM. Improving mental health in black men through a 24-week community-based lifestyle change intervention: the black impact program. BMC Psychiatry. 2024 Jan 9;24(1):34. doi: 10.1186/s12888-023-05064-5. PMID 38195473